CLINICAL TRIAL: NCT02899377
Title: A Pilot Study to Evaluate Molecular Imaging Methods in Primary Sjögren's Syndrome
Brief Title: A PH I Pilot Imaging Study to Evaluate Molecular Imaging Methods in HVs and pSS Pts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 203818
Record Dates: First submitted 2016-08-23; First posted 2016-09-14 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Autoimmune Diseases
Keywords: PET/CT; Primary Sjögren's Syndrome; Magnetic resonance imaging; 11^C-MET; 18^F-FDG
MeSH Terms: conditions — Autoimmune Diseases | interventions — gadoterate meglumine; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Health subjects (Experimental): During Visit 1, these subjects will undergo the following: An MRI of the salivary glands with one-time intravenous (IV) bolus injection of 0.1 mmol/kg of gadoterate meglumine and receive one-time IV bolus injection of 500 megabecquerels (MBq) of 11C MET followed by a PET/CT (dynamic scan of the salivary glands followed by head to hip static scan)
  Interventions: Radiation: 11C-MET PET/CT Imaging; Procedure: MRI Imaging with intravenous contrast with gadoterate meglumine
- Group B: pSS subjects (Experimental): During Visit 1, subjects with pSS will undergo the following: An MRI of the salivary glands with IV bolus injection of <=0.1 mmol/kg of gadoterate meglumine and receive one-time IV bolus injections: 500 MBq of 11C-MET (PET/CT: as for Group A) and 200 MBq of 18F-FDG followed by a PET/CT (static head to hip scan)
  Interventions: Radiation: 18F-FDG PET/CT Imaging; Radiation: 11C-MET PET/CT Imaging; Procedure: MRI Imaging with intravenous contrast with gadoterate meglumine; Procedure: Minor Salivary gland (labial) biopsy

INTERVENTIONS:
Radiation: 18F-FDG PET/CT Imaging — pSS subjects (in fasting conditions) will receive one-time bolus IV injection of 200 MBq of 18F-FDG. After 60 minutes of administration, a PET scan will be performed with static scanning acquired for up to 30 to 40 minutes.Other name: 18F-FDG
  Arms: Group B: pSS subjects
Radiation: 11C-MET PET/CT Imaging — Subjects (post meal) will receive one-time bolus IV injection of 500 MBq of 11C-MET. This will be followed by PET scan and dynamic scanning of the salivary gland region for approximately 40 minutes. A static scan will then be performed (within 5 minutes) with the whole body CT followed by the PET covering the head to hip with a duration of same range for approximately 20 to 30 minutes.
  Other Name:11C-MET
Procedure: MRI Imaging with intravenous contrast with gadoterate meglumine — Eligible subjects will receive a one-time IV injection of 0.1mmol/kg of gadoterate meglumine followed by a multi-parametric MRI scanning.
Procedure: Minor Salivary gland (labial) biopsy — A minor salivary gland biopsy will be performed at Visit 2 for pSS subjects only.
  Arms: Group B: pSS subjects

SUMMARY:
This is a pilot imaging study to determine whether molecular imaging with 18^F fluorodeoxyglucose (FDG) positron emission tomography (PET)/computed tomography (CT), 11^C-Methionine (MET) PET/CT, and salivary gland magnetic resonance imaging (MRI) with Dotarem (gadoterate meglumine) have the potential to characterize and quantify disease manifestations in primary Sjögren's syndrome (pSS) subjects. This will be achieved by assessing the associations and consistency between the imaging techniques studied, clinical assessments (salivary and tear flow and clinical scores), laboratory biomarkers, and histological findings on minor salivary gland biopsy.

In this study, healthy volunteers will be enrolled in Group A and pSS subjects in Group B. The subjects will be required to undergo screening and baseline assessments including unstimulated and stimulated salivary flow and Schirmer's test; an imaging visit (Visit 1); a sample collection visit (Visit 2) for repeat of selected baseline assessments and a minor salivary gland biopsy for pSS subjects only; and a follow-up visit. The total duration of participation in the study will be up to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* GROUP A: Healthy Volunteers Subjects for both PET/CT and MRI: Aged >=40 years inclusive at the time of signing the informed consent.

Subjects for MRI, without PET/CT: Aged >=30 years inclusive at the time of signing the informed consent Healthy as defined by the investigator, or medically qualified designee, based on a medical evaluation including medical history, physical examination, and laboratory tests.

* Group B: Primary Sjögren's Syndrome Patients Age >=30 years, at the time of signing the informed consent. Diagnosis of pSS according to the American-European Consensus Group criteria Baseline unstimulated salivary flow >0.0 mL/min or evidence of glandular reserve function (stimulated baseline salivary flow >0.05 mL/min).

Systemically active disease, ESSDAI >=5 points

* All Subjects Body weight >=50 kilogram (kg) and body mass index within the range 18.5 to 35 kg/m^2 (inclusive)

Male or Female, where one of the following conditions apply:

A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin test) at screening, and a negative urine pregnancy test 4-7 days prior to Visit 1, on the day of Visit 1 (on each day of scanning), on Visit 2, is not lactating, and at least one of the following conditions applies: non-reproductive potential or reproductive potential and agrees to use contraceptive methods listed in the protocol from 28 days prior to Visit 1 until follow up.

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form.

Exclusion Criteria:

* Diagnosis of secondary Sjögren's Syndrome.
* Diagnosis of another systemic autoimmune disease, apart from pSS, including but not limited to, systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis or systemic vasculitis. For Group B subjects, autoimmune conditions associated with pSS (for example autoimmune thyroiditis, primary biliary cirrhosis or coeliac disease), are not included in this exclusion, but should be described in the medical history taken baseline. If in doubt please consult the medical monitor.
* Subjects with active life-threatening or organ-threatening effects of pSS meaning that they may not be able to complete the study visits according to the protocol (as determine by the investigator) (Group B).
* History of coagulation or bleeding disorders which would increase the risk of minor salivary gland biopsy (for example, but not limited to, Hemophilia A or B, Von Willibrand's disease, platelet function disorders; Group B).
* History of malignancy within 5 years of screening that, in the view of the investigator, in consultation with the medical monitor if required, could confound the results of the 18F-FDG PET/CT scan (including lymphoma associated with pSS). This does not include cervical carcinoma in situ or non-melanoma skin malignancy that has been treated with curative surgical treatment.
* History of unresolved acute or chronic infection that, in the view of the investigator in consultation with the medial monitor, if required, could confound the results of the 18F-FDG PET/CT.
* Subject with diabetes mellitus requiring insulin therapy
* Contraindications to MRI scanning (as assessed by MRI safety questionnaire).
* History of, or suffers from, claustrophobia or feel that they will be unable to lie still in the PET or MRI scanner for a period of up to 1 to 2 hours.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* Previous inclusion in a research protocol involving nuclear medicine, PET or radiological investigations, or as a result of occupational exposure with a significant radiation burden (a significant radiation burden being defined as 10mSv in addition to natural background radiation, in the previous 3 years including the dose from this study). A clinical procedure where the subject received a direct benefit (eg diagnostic test) will not be included in the calculation of exposure.
* Lack of adequate peripheral venous access for cannulation.
* Current participation in a study with an investigational product, or recent participation within 5 half lives of discontinuation the drug, or within twice the duration of the biological effect of the drug, whichever is longer
* Group A: Healthy volunteers Subject is unable to refrain from taking prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 7 days prior to Visit 1 until completion of Visit 2, unless in the opinion of the investigator and Sponsor the medication will not interfere with the study.
* Group B: pSS subjects taking immunomodulatory treatment at screening are excluded unless they have been on stable doses of these medicines for 6 weeks prior to Screening/Baseline and are expected to remain on stable doses of these medications until the Follow up visit. This would include drugs such as glucocorticoids, immunosuppressive agents (for example, hydroxychloroquine, azathioprine, methotrexate, mycophenolate mofetil, and biologic therapies). If in doubt, to be discussed with the Medical Monitor.
* Group B: pSS subjects receiving treatment with anti-coagulant medications, including but not limited to warfarin, heparin, thrombin inhibitors, and Factor Xa inhibitors, and aspirin, unless the subjects is able to discontinue these medications one week prior to minor salivary gland biopsy, or according to local guidelines. The treatment may be restarted 3 days after the biopsy, or according to local guidelines.
* History of alcohol, prescription or non-prescription drug abuse which could interfere with participation in the trial according to the protocol, or in the opinion of the investigator impacts on the physical or mental wellbeing of the subject
* History of allergy/hypersensitivity to study medications including local anesthesia (Group B), radio-isotopes or gadolinium-containing contrast agents (all subjects).
* Contraindications to gadolinium-containing contrast agents in accordance with product labeling and local guidelines
* Estimated GFR (Modification of Diet in Renal Disease calculation) of less than 60 mL/min/1.73m^2 at screening.
* Platelet count below the laboratory normal range at screening, or prothrombin time above the laboratory normal range at screening (Group B).
* Subject with a fasting blood sugar >11.1 millimoles (mmol)/Liters (L) at screening (defined as fasting for a minimum of 6 hours, excluding unflavored water).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a pilot imaging study using positron emission tomography (PET)/computed tomography (CT) and multi parametric magnetic resonance imaging (MRI) to investigate the potential to characterize and quantify disease manifestation in primary Sjögren's syndrome (pSS) participants.
Pre-assignment Details: A total of 25 participants were enrolled in the study. The study was conducted at 3 centers in the United Kingdom.
Groups:
- Healthy Participants: Underwent an MRI of the salivary glands with one-time intravenous (IV) bolus injection of 0.1 millimoles (mmol)/kilogram (kg) of gadoterate meglumine and received one-time IV bolus injection of 500 megabecquerels (MBq) of carbon11-methionine (11C -MET) followed by a PET/CT (dynamic scan of the salivary glands followed by head to hip static scan)
- Participants With pSS: Underwent an MRI of the salivary glands with IV bolus injection of <=0.1 mmol/kg of gadoterate meglumine and received one-time IV bolus injections: 500 MBq of 11C-MET and 200 MBq of 18F-flurodeoxyglucose (FDG) followed by a PET/CT (static head to hip scan).
Period: Overall Study
Arm/Group | Healthy Participants | Participants With pSS
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Participants: Underwent an MRI of the salivary glands with one-time IV bolus injection of 0.1 mmol/kg of gadoterate meglumine and received one-time IV bolus injection of 500 MBq of 11C-MET followed by a PET/CT (dynamic scan of the salivary glands followed by head to hip static scan)
- Participants With pSS: Underwent an MRI of the salivary glands with IV bolus injection of <=0.1 mmol/kg of gadoterate meglumine and received one-time IV bolus injections: 500 MBq of 11C-MET and 200 MBq of 18F-FDG followed by a PET/CT (static head to hip scan).
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Participants With pSS | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (13.87) | 49.0 (13.70) | 48.5 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian: Central/south Asian heritage | 0 | 3 | 3
  Asian: South East Asian heritage | 0 | 1 | 1
  Black or African American | 2 | 0 | 2
  White/Caucasian/European Heritage | 10 | 5 | 15
  Mixed race White Caribbean | 1 | 0 | 1
  Unknown | 0 | 2 | 2
  Black British | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Standardized Uptake Value (SUV) for 18F-FDG for pSS Participants in Selected Body Areas
Description: Semi-quantitative parameters used for the assessment of glucose uptake included Mean, Peak and Max SUV for following selected body areas: aorta, liver, muscle, pancreas, lumbar vertebra, salivary gland, spleen, and thyroid. Safety Population included all participants who underwent any procedure on or after Visit 1.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Participants With pSS
Number analyzed (Participants) | 12
Grams per milliliter
  Aorta, Max SUV | 2.9067 (0.49445)
  Liver, Max SUV | 5.0683 (1.13564)
  Lumbar Vertebra, Max SUV | 4.0225 (0.91105)
  Muscle, Max SUV | 1.4558 (0.50282)
  Pancreas, Max SUV | 4.2700 (1.02711)
  Salivary gland, Max SUV | 3.1067 (0.83496)
  Spleen, Max SUV | 3.2333 (0.54135)
  Thyroid, Max SUV | 3.1408 (0.72742)
  Aorta, Mean SUV | 1.883 (0.2740)
  Liver, Mean SUV | 2.273 (0.2605)
  Lumbar Vertebra, Mean SUV | 2.105 (0.4000)
  Muscle, Mean SUV | 0.657 (0.1696)
  Pancreas, Mean SUV | 1.874 (0.2511)
  Spleen, Mean SUV | 1.751 (0.1889)
  Thyroid, Mean SUV | 1.822 (0.5509)
  Aorta, Peak SUV | 2.0125 (0.35028)
  Liver, Peak SUV | 3.2700 (0.53533)
  Lumbar Vertebra, Peak SUV | 2.8242 (0.58906)
  Muscle, Peak SUV | 0.8833 (0.25378)
  Pancreas, Peak SUV | 2.6892 (0.47389)
  Salivary gland, Peak SUV | 2.1425 (0.58856)
  Spleen, Peak SUV | 2.3475 (0.30266)
  Thyroid, Peak SUV | 2.2458 (0.68193)

2. Primary Outcome: SUV of Lachrymal Gland, Parotid Gland, and Submandibular Gland for 18F-FDG for pSS Participants
Description: Semi-quantitative parameters used for the assessment of glucose uptake included Mean, Peak and Max SUV for following selected body areas: lachrymal gland, parotid gland, and submandibular gland. Data for lower value of region (low), higher value of region (high), and aggregated value which is left and right region combined value has been reported for the regions of interest. SUV is a mathematically derived ratio of tissue radioactivity concentration and the injected dose of radioactivity per kilogram of the participant's body weight at a given point in time.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Participants With pSS
Number analyzed (Participants) | 12
Grams per milliliter
  Lachrymal gland, Low, Max SUV | 1.7808 (0.38311)
  Lachrymal gland, High, Max SUV | 2.0658 (0.34849)
  Lachrymal gland, Aggregated, Max SUV | 2.0658 (0.34849)
  Parotid gland, Low, Max SUV | 2.5767 (0.68672)
  Parotid gland, High, Max SUV | 2.7783 (0.76902)
  Parotid gland, Aggregated, Max SUV | 2.7783 (0.76902)
  Submandibular gland, Low, Max SUV | 2.5200 (0.82131)
  Submandibular gland, High, Max SUV | 2.9250 (0.94362)
  Submandibular gland, Aggregated, Max SUV | 2.9250 (0.94362)
  Lachrymal gland, Low, Mean SUV | 1.311 (0.3218)
  Lachrymal gland, High, Mean SUV | 1.515 (0.2934)
  Parotid gland, Low, Mean SUV | 1.620 (0.5022)
  Parotid gland, High, Mean SUV | 1.818 (0.5957)
  Submandibular gland, Low, Mean SUV | 1.709 (0.6786)
  Submandibular gland, High, Mean SUV | 1.916 (0.6237)
  Lachrymal gland, Low, Peak SUV | 1.5842 (0.18535)
  Lachrymal gland, High, Peak SUV | 1.7125 (0.24264)
  Lachrymal gland, Aggregated, Peak SUV | 1.6492 (0.20505)
  Parotid gland, Low, Peak SUV | 2.0150 (0.64590)
  Parotid gland, High, Peak SUV | 2.2383 (0.71837)
  Parotid gland, Aggregated, Peak SUV | 2.1275 (0.67216)
  Submandibular gland, Low, Peak SUV | 1.9275 (0.74620)
  Submandibular gland, High, Peak SUV | 2.3883 (0.69049)
  Submandibular gland, Aggregated, Peak SUV | 2.1583 (0.67168)

3. Primary Outcome: Tissue to Reference (TR) Ratio for 18F- FDG for pSS Participants
Description: Semi-quantitative parameters used for the assessment of glucose uptake included TR ratio for the following selected body areas: aorta, liver, lumbar vertebra, muscle, pancreas, salivary gland, spleen, and thyroid.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Participants With pSS
Number analyzed (Participants) | 12
Ratio
  Aorta | 1.0660 (0.05729)
  Liver | 1.7366 (0.11645)
  Lumbar Vertebra | 1.5096 (0.28568)
  Muscle | 0.4669 (0.10222)
  Pancreas | 1.4312 (0.16490)
  Salivary gland | 1.1730 (0.38592)
  Spleen | 1.2625 (0.17400)
  Thyroid | 1.2193 (0.44934)

4. Primary Outcome: TR Ratio of Lachrymal Gland, Parotid Gland, and Submandibular Gland for 18F-FDG for pSS Participants
Description: Semi-quantitative parameters used for the assessment of glucose uptake included TR ratio for following selected body areas: lachrymal gland, parotid gland, and submandibular gland. Data for lower value of region (low), higher value of region (high), and aggregated value which includes left and right region combined value has been reported.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Participants With pSS
Number analyzed (Participants) | 12
Ratio
  Lachrymal gland, Low | 0.8529 (0.12250)
  Lachrymal gland, High | 0.9201 (0.13587)
  Lachrymal gland, Aggregated | 0.8864 (0.12560)
  Parotid gland, Low | 1.1158 (0.44262)
  Parotid gland, High | 1.2338 (0.47055)
  Parotid gland, Aggregated | 1.1749 (0.45273)
  Submandibular gland, Low | 1.0472 (0.43105)
  Submandibular gland, High | 1.2953 (0.41063)
  Submandibular gland, Aggregated | 1.1711 (0.40012)

5. Primary Outcome: Total Inflammatory Volume for 18F- FDG for pSS Participants at Selected Body Areas
Description: There were no anatomically relevant areas indicative of inflamed tissue and/or focal uptake within the organs that would warrant calculation of TIV
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population. Data was not collected
Arm/Group | Participants With pSS
Number analyzed (Participants) | 0

6. Primary Outcome: SUV for 11C- MET in Selected Body Areas
Description: Semi-quantitative parameters used for the assessment of uptake included Mean, Peak and Max SUV for following selected body areas: aorta, liver, muscle, lumbar vertebra, pancreas, salivary gland, spleen, and thyroid. Data from static scan is reported.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Participants With pSS | Healthy Participants
Number analyzed (Participants) | 12 | 8
Grams per milliliter
  Aorta, Max SUV | 2.2700 (0.72709) | 2.0275 (0.62609)
  Liver, Max SUV | 19.1667 (3.81783) | 16.4213 (3.31237)
  Lumbar Vertebra, Max SUV | 7.1733 (2.85382) | 5.9100 (1.43376)
  Muscle, Max SUV | 2.4167 (0.89879) | 2.3513 (1.01454)
  Pancreas, Max SUV | 31.4492 (5.17911) | 31.7388 (5.68871)
  Salivary gland, Max SUV | 5.4275 (1.43053) | 6.6900 (1.05224)
  Spleen, Max SUV | 5.5100 (1.35700) | 5.2750 (1.22413)
  Thyroid, Max SUV | 3.7058 (0.86450) | 3.1038 (0.79784)
  Aorta, Mean SUV | 1.161 (0.2927) | 1.029 (0.3334)
  Liver, Mean SUV | 10.926 (2.1692) | 8.916 (1.4380)
  Lumbar Vertebra, Mean SUV | 3.485 (0.9351) | 2.923 (0.5387)
  Muscle, Mean SUV | 0.968 (0.2074) | 0.926 (0.2365)
  Pancreas, Mean SUV | 16.413 (3.1008) | 16.556 (2.9023)
  Spleen, Mean SUV | 2.650 (0.3745) | 2.423 (0.1005)
  Thyroid, Mean SUV | 2.149 (0.6418) | 1.646 (0.3138)
  Aorta, Peak SUV | 1.3250 (0.37590) | 1.1338 (0.41008)
  Liver, Peak SUV | 14.7808 (3.01666) | 12.3438 (1.76812)
  Lumbar Vertebra, Peak SUV | 4.7317 (1.28105) | 3.8775 (0.62923)
  Muscle, Peak SUV | 1.3675 (0.40656) | 1.3100 (0.29544)
  Pancreas, Peak SUV | 26.4683 (4.29608) | 26.7913 (6.21700)
  Salivary gland, Peak SUV | 3.3633 (1.16624) | 5.0600 (0.83111)
  Spleen, Peak SUV | 3.6975 (0.61556) | 3.4100 (0.35633)
  Thyroid, Peak SUV | 2.6000 (0.65448) | 2.0525 (0.29673)

7. Primary Outcome: SUV of Lachrymal Gland, Parotid Gland, and Submandibular Gland for 11C-MET
Description: Semi-quantitative parameters used for the assessment of uptake included Mean, Peak and Max SUV for following selected body areas: lachrymal gland, parotid gland, and submandibular gland. Data from static scan for lower value of region (low), higher value of region (high), and aggregated value which includes left and right region combined value has been reported. SUV is a mathematically derived ratio of tissue radioactivity concentration and the injected dose of radioactivity per kilogram of the participant's body weight at a given point in time.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Grams per milliliter
Arm/Group | Participants With pSS | Healthy Participants
Number analyzed (Participants) | 12 | 8
Grams per milliliter
  Lachrymal gland, Low, Max SUV | 1.9133 (1.00469) | 2.5513 (1.00049)
  Lachrymal gland, High, Max SUV | 2.1483 (1.02205) | 3.1250 (1.49196)
  Lachrymal gland, Aggregated, Max SUV | 2.1483 (1.02205) | 3.1250 (1.49196)
  Parotid gland, Low, Max SUV | 4.3933 (1.31072) | 5.9038 (1.01547)
  Parotid gland, High, Max SUV | 4.9492 (1.22415) | 6.3750 (1.09929)
  Parotid gland, Aggregated, Max SUV | 4.9492 (1.22415) | 6.3750 (1.09929)
  Submandibular gland, Low, Max SUV | 3.8583 (1.78484) | 6.2150 (1.06158)
  Submandibular gland, High, Max SUV | 4.4692 (1.77872) | 6.5488 (0.94266)
  Submandibular gland, Aggregated, Max SUV | 4.4692 (1.77872) | 6.5488 (0.94266)
  Lachrymal gland, Low, Mean SUV | 1.312 (0.6048) | 1.703 (0.5810)
  Lachrymal gland, High, Mean SUV | 1.462 (0.6490) | 2.056 (0.7874)
  Parotid gland, Low, Mean SUV | 2.525 (0.8740) | 3.505 (0.5637)
  Parotid gland, High, Mean SUV | 2.925 (0.8679) | 3.648 (0.5709)
  Submandibular gland, Low, Mean SUV | 2.388 (1.1855) | 3.923 (0.4941)
  Submandibular gland, High, Mean SUV | 2.648 (1.2128) | 4.191 (0.5410)
  Lachrymal gland, Low, Peak SUV | 1.3525 (0.59715) | 1.7738 (0.66125)
  Lachrymal gland, High, Peak SUV | 1.4958 (0.65626) | 2.1688 (0.99580)
  Lachrymal gland, Aggregated, Peak SUV | 1.4233 (0.62222) | 1.9713 (0.81354)
  Parotid gland, Low, Peak SUV | 3.4367 (1.22748) | 4.9000 (0.92893)
  Parotid gland, High, Peak SUV | 3.9175 (1.18255) | 5.1663 (0.85276)
  Parotid gland, Aggregated, Peak SUV | 3.6767 (1.18792) | 5.0325 (0.89020)
  Submandibular gland, Low, Peak SUV | 2.8025 (1.53196) | 4.8588 (0.86087)
  Submandibular gland, High, Peak SUV | 3.2992 (1.63167) | 5.3100 (0.89113)
  Submandibular gland, Aggregated, Peak SUV | 3.0517 (1.56359) | 5.0838 (0.86490)

8. Primary Outcome: TR Ratio for 11C- MET
Description: Semi-quantitative parameters used for the assessment of uptake included TR ratio for following selected body areas: aorta, liver, muscle, lumbar vertebra, pancreas, salivary gland, spleen, and thyroid. Data from static scan has been reported.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Participants With pSS | Healthy Participants
Number analyzed (Participants) | 12 | 8
Ratio
  Aorta | 1.1352 (0.06738) | 1.0910 (0.04942)
  Liver | 13.1513 (3.13572) | 12.8649 (3.46136)
  Lumbar Vertebra | 4.1158 (0.85314) | 3.9731 (0.80867)
  Muscle | 1.1914 (0.26802) | 1.3354 (0.34831)
  Pancreas | 23.5403 (4.62140) | 29.8331 (15.21426)
  Salivary gland | 3.0974 (1.30105) | 5.2805 (1.44642)
  Spleen | 3.2872 (0.67470) | 3.5414 (0.81253)
  Thyroid | 2.3002 (0.63142) | 2.1213 (0.49670)

9. Primary Outcome: TR Ratio for 11C- MET of Salivary Glands, Lachrymal Gland, Parotid Gland, and Submandibular Gland
Description: Semi-quantitative parameters used for the assessment of uptake included TR ratio for following selected body areas: lachrymal gland, parotid gland, and submandibular gland. Data from static scan for lower value of region (low), higher value of region (high), and aggregated value which includes left and right region combined value has been reported.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Participants With pSS | Healthy Participants
Number analyzed (Participants) | 12 | 8
Ratio
  Lachrymal gland, Low | 1.2007 (0.55639) | 1.8219 (0.62711)
  Lachrymal gland, High | 1.3178 (0.59115) | 2.1965 (0.76588)
  Lachrymal gland, Aggregated | 1.2594 (0.57188) | 2.0094 (0.68084)
  Parotid gland, Low | 3.1810 (1.44525) | 5.1570 (1.61371)
  Parotid gland, High | 3.6198 (1.41338) | 5.4621 (1.73285)
  Parotid gland, Aggregated | 3.4003 (1.41542) | 5.3096 (1.67006)
  Submandibular gland, Low | 2.5766 (1.61682) | 5.0230 (1.20994)
  Submandibular gland, High | 3.0126 (1.61982) | 5.4796 (1.30126)
  Submandibular gland, Aggregated | 2.7946 (1.60578) | 5.2513 (1.24653)

10. Primary Outcome: Total Inflammatory Volume 11C- MET at Selected Body Areas
Description: as for outcome 5
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population. Data was not collected
Arm/Group | Participants With pSS | Healthy Participants
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Multi-parametric MRI Derived Parameter: Apparent Diffusion Coefficient (ADC)
Description: Quantitative parameters like ADC assessed use of multi-parametric MRI in the assessment of uptake in selected body areas like lachrymal gland, parotid gland, and submandibular gland. The median and interquartile range (IQR) values for ADC was used for analysis. Data for lower value of region (low), higher value of region (high), and aggregated value which includes left and right region combined value has been reported.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Error); unit: 10^-3 square millimeter per second
Arm/Group | Healthy Participants | Participants With pSS
Number analyzed (Participants) | 13 | 12
10^-3 square millimeter per second
  Parotid Gland, Low, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Low, IQR, n=12, 11 | 0.511 (0.0314) | 0.516 (0.0356)
  Parotid Gland, High, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, High, IQR, n=12, 11 | 0.581 (0.0275) | 0.646 (0.0412)
  Parotid Gland, Aggregated, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Aggregated, IQR, n=12, 11 | 0.544 (0.0264) | 0.582 (0.0408)
  Submandibular Gland, Low, IQR, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, Low, IQR, n=12, 10 | 0.549 (0.0321) | 0.765 (0.0693)
  Submandibular Gland, High, IQR, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, High, IQR, n=12, 10 | 0.674 (0.0309) | 0.928 (0.0714)
  Submandibular Gland, Aggregated, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Submandibular Gland, Aggregated, IQR, n=12, 11 | 0.602 (0.0303) | 0.809 (0.0695)
  Parotid Gland, Low, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Low, Median, n=12, 11 | 1.091 (0.0476) | 1.011 (0.0607)
  Parotid Gland, High, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, High, Median, n=12, 11 | 1.153 (0.0451) | 1.117 (0.0524)
  Parotid Gland, Aggregated, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Aggregated, Median, n=12, 11 | 1.120 (0.0460) | 1.069 (0.0539)
  Submandibular Gland, Low, Median, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, Low, Median, n=12, 10 | 1.469 (0.0377) | 1.410 (0.0924)
  Submandibular Gland, High, Median, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, High, Median, n=12, 10 | 1.540 (0.0461) | 1.551 (0.0833)
  Submandibular Gland, Aggregated, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Submandibular Gland, Aggregated, Median, n=12, 11 | 1.506 (0.0396) | 1.474 (0.0767)

12. Primary Outcome: Multi-parametric MRI Derived Parameter: Pure Diffusion Coefficient (D)
Description: Quantitative parameters like pure D assessed the use of multi-parametric MRI in the assessment of uptake in selected body areas like lachrymal gland, parotid gland, and submandibular gland. The median and IQR values for pure D was used for analysis. Data for lower value of region, higher value of region, and aggregated value which includes left and right region combined value has been reported.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: as for outcome 11
Measure: Mean (Standard Error); unit: 10^-3 square millimeter per second
Arm/Group | Healthy Participants | Participants With pSS
Number analyzed (Participants) | 13 | 12
10^-3 square millimeter per second
  Parotid Gland, Low, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Low, IQR, n=12, 11 | 0.437 (0.0343) | 0.449 (0.0326)
  Parotid Gland, High, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, High, IQR, n=12, 11 | 0.503 (0.0336) | 0.529 (0.0296)
  Parotid Gland, Aggregated, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Aggregated, IQR, n=12, 11 | 0.468 (0.0344) | 0.493 (0.0322)
  Submandibular Gland, Low, IQR, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, Low, IQR, n=12, 10 | 0.553 (0.0361) | 0.547 (0.0440)
  Submandibular Gland, High, IQR, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, High, IQR, n=12, 10 | 0.733 (0.0377) | 0.681 (0.0641)
  Submandibular Gland, Aggregated, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Submandibular Gland, Aggregated, IQR, n=12, 11 | 0.636 (0.0324) | 0.608 (0.0443)
  Parotid Gland, Low, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Low, Median, n=12, 11 | 0.771 (0.0269) | 0.621 (0.0492)
  Parotid Gland, High, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, High, Median, n=12, 11 | 0.807 (0.0287) | 0.715 (0.0450)
  Parotid Gland, Aggregated, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Aggregated, Median, n=12, 11 | 0.787 (0.0274) | 0.676 (0.0457)
  Submandibular Gland, Low, Median, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, Low, Median, n=12, 10 | 0.941 (0.0445) | 0.733 (0.0924)
  Submandibular Gland, High, Median, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, High, Median, n=12, 10 | 1.035 (0.0402) | 0.814 (0.0887)
  Submandibular Gland, Aggregated, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Submandibular Gland, Aggregated, Median, n=12, 11 | 0.993 (0.0409) | 0.807 (0.0905)

13. Primary Outcome: Multi-parametric MRI Derived Parameter: Microvascular Volume Fraction
Description: Quantitative parameters like Microvascular Volume Fraction assessed use of multi-parametric MRI in selected body areas like lachrymal gland, parotid gland, and submandibular gland. The median and IQR values were used for analysis. Data for lower value of region, higher value of region, and aggregated value which includes left and right region combined value has been reported. The IVIM (intra-voxel incoherent motion) model estimates two separate pools of diffusion (for a microvascular component and a tissue component). Pool one describes fraction (f) of the signal. Pool two describes fraction (1-f) of the signal. Microvascular Volume Fraction (f) is the ratio of the signal contribution of the microvascular pool (pool one) over the entire signal.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: as for outcome 11
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Healthy Participants | Participants With pSS
Number analyzed (Participants) | 13 | 12
Ratio
  Parotid Gland, Low, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Low, IQR, n=12, 11 | 0.135 (0.0084) | 0.135 (0.0122)
  Parotid Gland, High, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, High, IQR, n=12, 11 | 0.164 (0.0082) | 0.172 (0.0155)
  Parotid Gland, Aggregated, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Aggregated, IQR, n=12, 11 | 0.149 (0.0090) | 0.156 (0.0145)
  Submandibular Gland, Low, IQR, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, Low, IQR, n=12, 10 | 0.204 (0.0126) | 0.205 (0.0101)
  Submandibular Gland, High, IQR, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, High, IQR, n=12, 10 | 0.233 (0.0143) | 0.233 (0.0102)
  Submandibular Gland, Aggregated, IQR, n=12, 11: number analyzed (Participants) | 12 | 11
  Submandibular Gland, Aggregated, IQR, n=12, 11 | 0.219 (0.0135) | 0.217 (0.0097)
  Parotid Gland, Low, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Low, Median, n=12, 11 | 0.131 (0.0068) | 0.139 (0.0068)
  Parotid Gland, High, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, High, Median, n=12, 11 | 0.151 (0.0098) | 0.164 (0.0127)
  Parotid Gland, Aggregated, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Parotid Gland, Aggregated, Median, n=12, 11 | 0.140 (0.0079) | 0.151 (0.0100)
  Submandibular Gland, Low, Median, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, Low, Median, n=12, 10 | 0.198 (0.0164) | 0.238 (0.0263)
  Submandibular Gland, High, Median, n=12, 10: number analyzed (Participants) | 12 | 10
  Submandibular Gland, High, Median, n=12, 10 | 0.223 (0.0167) | 0.271 (0.0257)
  Submandibular Gland, Aggregated, Median, n=12, 11: number analyzed (Participants) | 12 | 11
  Submandibular Gland, Aggregated, Median, n=12, 11 | 0.210 (0.0165) | 0.243 (0.0273)

14. Primary Outcome: Multi-parametric MRI Derived Parameter: Exchange Rate (KTrans)
Description: Quantitative parameters like KTrans assessed use of multi-parametric MRI in the assessment of uptake in selected body areas like lachrymal gland, parotid gland, and submandibular gland. The median and IQR values were used for analysis. Data for lower value of region, higher value of region, and aggregated value which includes left and right region combined value has been reported.
Time Frame: Visit 1: Within 6 weeks after Baseline
Population: as for outcome 11
Measure: Mean (Standard Error); unit: Per minute
Arm/Group | Healthy Participants | Participants With pSS
Number analyzed (Participants) | 13 | 12
Per minute
  Parotid Gland, Low, IQR, n=12, 12: number analyzed (Participants) | 12 | 12
  Parotid Gland, Low, IQR, n=12, 12 | 7.618 (3.8286) | 22.492 (9.8803)
  Parotid Gland, High, IQR, n=12, 12: number analyzed (Participants) | 12 | 12
  Parotid Gland, High, IQR, n=12, 12 | 12.821 (6.7497) | 30.199 (13.2411)
  Parotid Gland, Aggregated, IQR, n=12, 12: number analyzed (Participants) | 12 | 12
  Parotid Gland, Aggregated, IQR, n=12, 12 | 10.701 (5.5677) | 27.213 (12.3396)
  Submandibular Gland, Low, IQR, n=9, 8: number analyzed (Participants) | 9 | 8
  Submandibular Gland, Low, IQR, n=9, 8 | 5.548 (4.6510) | 0.459 (0.0850)
  Submandibular Gland, High, IQR, n=9, 8: number analyzed (Participants) | 9 | 8
  Submandibular Gland, High, IQR, n=9, 8 | 15.192 (9.3625) | 19.914 (17.5121)
  Submandibular Gland, Aggregated, IQR, n=11, 11: number analyzed (Participants) | 11 | 11
  Submandibular Gland, Aggregated, IQR, n=11, 11 | 10.191 (6.1313) | 1.801 (0.8246)
  Parotid Gland, Low, Median, n=12, 12: number analyzed (Participants) | 12 | 12
  Parotid Gland, Low, Median, n=12, 12 | 5.598 (2.5910) | 3.326 (1.3677)
  Parotid Gland, High, Median, n=12, 12: number analyzed (Participants) | 12 | 12
  Parotid Gland, High, Median, n=12, 12 | 8.841 (4.3542) | 9.323 (4.9569)
  Parotid Gland, Aggregated, Median, n=12, 12: number analyzed (Participants) | 12 | 12
  Parotid Gland, Aggregated, Median, n=12, 12 | 7.061 (3.4227) | 7.450 (3.8203)
  Submandibular Gland, Low, Median, n=9, 8: number analyzed (Participants) | 9 | 8
  Submandibular Gland, Low, Median, n=9, 8 | 12.789 (11.7785) | 0.775 (0.2742)
  Submandibular Gland, High, Median, n=9, 8: number analyzed (Participants) | 9 | 8
  Submandibular Gland, High, Median, n=9, 8 | 17.315 (12.2640) | 1.606 (0.5826)
  Submandibular Gland, Aggregated, Median, n=11,11: number analyzed (Participants) | 11 | 11
  Submandibular Gland, Aggregated, Median, n=11,11 | 12.146 (9.8325) | 1.421 (0.6603)

15. Secondary Outcome: Net Irreversible Influx Rate Constant (Ki) From 11C-MET PET/CT
Description: Blood samples were collected at indicated time points for radio-pharmacokinetic analysis of Ki. Pharmacokinetic (PK) Population included those participants in the 'Safety' population for whom a radio-pharmacokinetic sample was obtained and analyzed. Data for lower value of region (low), higher value of region (high) and right-left combined values (aggregated) is presented.
Time Frame: 0.1, 0.4, 0.6, 0.9, 1.1, 1.4, 1.6, 1.9, 2.5, 3.5, 4.5, 6.0, 8, 10, 12, 14, 17.5, 22.5, 27.5, 32.5 and 37.5 minutes post-injection
Population: PK Population
Measure: Mean (Standard Deviation); unit: Milliliter/centimeter cube/minute
Arm/Group | Healthy Participants | Participants With pSS
Number analyzed (Participants) | 8 | 12
Milliliter/centimeter cube/minute
  Parotid Gland, Low | 0.0574 (0.02282) | 0.0425 (0.02200)
  Parotid Gland, High | 0.0608 (0.02411) | 0.0472 (0.02293)
  Parotid Gland, Aggregated | 0.0593 (0.02332) | 0.0448 (0.02211)
  Submandibular Gland, Low | 0.0598 (0.02051) | 0.0383 (0.01756)
  Submandibular Gland, High | 0.0626 (0.02137) | 0.0422 (0.01916)
  Submandibular Gland, Aggregated | 0.0614 (0.02085) | 0.0407 (0.01863)

16. Secondary Outcome: Correlation Between Static and Dynamic Imaging Metrics in 11C-MET
Description: Blood samples were collected at indicated time points for analysis. Pearson's correlation is presented along with 95% confidence interval.
Time Frame: as for outcome 15
Population: PK Population
Measure: Number (95% Confidence Interval); unit: Grams per milliliter
Arm/Group | Healthy Participants | Participants With pSS
Number analyzed (Participants) | 8 | 12
Grams per milliliter
  Max SUV, Low | -0.066 [-0.736 to 0.670] | 0.915 [0.719 to 0.976]
  Max SUV, High | -0.106 [-0.754 to 0.647] | 0.884 [0.629 to 0.967]
  Max SUV, Aggregated | -0.100 [-0.752 to 0.650] | 0.891 [0.648 to 0.969]
  Mean SUV, Low | 0.142 [-0.625 to 0.770] | 0.895 [0.660 to 0.970]
  Mean SUV, High | 0.130 [-0.633 to 0.764] | 0.786 [0.387 to 0.937]
  Peak SUV, Low | 0.045 [-0.681 to 0.727] | 0.929 [0.761 to 0.980]
  Peak SUV, High | 0.053 [-0.677 to 0.730] | 0.866 [0.582 to 0.962]
  Peak SUV, Aggregated | 0.038 [-0.685 to 0.723] | 0.906 [0.692 to 0.974]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events and serious adverse events (SAE) were collected up to 11 weeks
Description: Non-serious adverse events and SAEs were collected for Safety Population
Arm/Group | Healthy Participants | Participants With pSS
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 1/13 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Participants (N=13) | Participants With pSS (N=12)
Headache (Nervous system disorders) | 1 (1) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT02899377/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02899377/SAP_001.pdf